CLINICAL TRIAL: NCT02118311
Title: T Regulatory Cell for Suppression of Acute Graft-vs-Host-Disease in Recipients of a Non-Myeloablative Umbilical Cord Blood Transplantation for Treatment of Hematological Malignancies
Brief Title: Treg Cells for AGVHD in Non-myeloablative UCB Transplant
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Changing study design. Will replace with a different protocol.
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013LS091; MT2013-27 (Other: University of Minnesota Blood and Marrow Transplant Program); P01CA065493 (NIH)
Record Dates: First submitted 2014-03-26; First posted 2014-04-21 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Hematologic Malignancies
Keywords: Acute Leukemias; Burkitt's Lymphoma; Natural Killer Cell Malignancies; Chronic Myelogenous Leukemia; Myelodysplastic Syndrome; Large-Cell Lymphoma; Hodgkin Lymphoma; Multiple Myeloma; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Marginal Zone B-Cell Lymphoma; Follicular Lymphoma:; Lymphoplasmacytic Lymphoma; Mantle-Cell Lymphoma; Prolymphocytic Leukemia
MeSH Terms: conditions — Hematologic Neoplasms; Burkitt Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Dendritic Cell Sarcoma, Interdigitating; Hodgkin Disease; Multiple Myeloma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Prolymphocytic | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TREG (Experimental): T regulatory cells after non-myeloablative (using fludarabine, cyclophosphamide, and total body irradiation) umbilical cord transplant.
  Interventions: Biological: T Regulatory cells; Drug: Fludarabine; Drug: Cyclophosphamide; Radiation: Total Body Irradiation
- Non-Myeloablative Only (Experimental): Non-myeloablative (using fludarabine, cyclophosphamide, and total body irradiation) umbilical cord transplant.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Radiation: Total Body Irradiation

INTERVENTIONS:
Biological: T Regulatory cells — Fixed dose of nTreg cells will be infused on day 0 of transplant after the umbilical cord blood cells
  Other Names: nTreg; Treg
  Arms: TREG
Drug: Fludarabine — Fludarabine 30mg/m^2 IV over 1 hour on days -6 through -2 from transplant
  Other Names: Fludara
Drug: Cyclophosphamide — Cyclophosphamide 50 mg/kg IV over 2 hours on day -6 from transplant
  Other Names: Endoxan; Cytoxan; Neosar; Procytox; Revimmune
Radiation: Total Body Irradiation — Total Body Irradiation (TBI) 200 cGy administered on day -1 in a single fraction will be given at a dose rate of 10-19 cGy/minute prescribed to the midplane of the patient at the level of the umbilicus.
  Other Names: TBI

SUMMARY:
This is a Simon's optimal two-stage phase II trial designed to estimate grade II-IV acute graft-versus-host disease (GVHD) after infusion of T regulatory (nTreg) in a fixed dose ratio to the combined CD3+ cell count of the two graft units in recipients of double UCB transplantation. The nTreg cells (manufactured from a 3rd cord blood unit) are infused on day 0 at least 1 hour after the 2nd unit of the double umbilical cord blood (UCB) transplant.

The nTreg cells require an 18 day (±2 days) lead time based on the planned transplant day. The combined CD3+ cell content from the two graft UCB units is enumerated upon thaw (day 0). The patient then receives the number of nTregs cells from the 3rd cord product to achieve a Treg:CD3+ cells ratio of 5:1. The nTreg cell dose depends on the CD3+ cell content of the two graft UCB graft units, but it will not exceed the highest dose level safely tested in the ongoing University of Minnesota phase I Treg dose escalation study MT 2006-01.

ELIGIBILITY:
Inclusion Criteria:

* Must be ≥18, but < 70 years of age with no matched 5/6 or 6/6 sibling donor - patients ≥ 70 and ≤ 75 years of age may be eligible if they have a Co-Morbidity score ≤ 2 (Appendix II)
* Three UCB units composing the graft will be selected according to the current University of Minnesota umbilical cord blood graft selection algorithm.
* Each UCB unit must be matched at 4-6 HLA-A, B, DRB1 antigens with the recipient. This may include 0-2 antigen mismatches at the A or B or DRB1 loci. Each unit must be a 4-6 HLA-A, B, DRB1 antigen match to each other, not necessarily at the same loci they are matched to the recipient.
* Disease Criteria

  * Acute Leukemias: Must be in remission by morphology (<5% blasts). Note cytogenetic relapse or persistent disease without morphologic relapse is acceptable. Also a small percentage of blasts that is equivocal between marrow regeneration versus early relapse are acceptable provided there are no associated cytogenetic markers consistent with relapse.
* Acute Lymphoblastic Leukemia (ALL) in first complete remission (CR1) that is NOT considered favorable-risk as defined by the presence of at least one of the following:

  * Adverse cytogenetics such as t(9;22), t(1;19), t(4;11), other MLL rearrangements
  * White blood cell counts of greater than 30,000/mcL (B-ALL) or greater than 100,000/mcL (T-ALL) at diagnosis
  * Recipient age older than 30 years at diagnosis
  * Time to CR greater than 4 weeks
* Acute Myelogenous Leukemia (AML) in first complete remission (CR1) that is NOT considered as favorable-risk. Favorable risk is defined as having one of the following:

  * t(8,21) without CKIT mutation
  * inv(16) without CKIT mutation or t(16;16)
  * Normal karyotype with mutated NPM1 and not FLT-IND
  * Normal karyotype with double mutated CEBPA
  * APL in first molecular remission at end of consolidation
* Acute Leukemias in 2nd or subsequent CR
* Biphenotypic/Undifferentiated in first or subsequent CR, adult T-cell leukemia/lymphoma in first or subsequent complete remission (CR)

  * Burkitt's Lymphoma in CR2 or subsequent complete remission (CR)
  * Natural Killer Cell Malignancies
  * Chronic Myelogenous Leukemia: all types except refractory blast crisis. Chronic phase patients must have failed or been intolerant to at least one tyrosine-kinase inhibitor
  * Myelodysplastic Syndrome: any subtype including refractory anemia (RA) if severe pancytopenia or complex cytogenetics. Blasts must be less than 5%. If 5% or more requires induction therapy pre-transplant to reduce blast count to ≤5%.
  * Large-Cell Lymphoma, Hodgkin Lymphoma and Multiple Myeloma with chemotherapy sensitive disease that has failed or patients who are ineligible for an autologous transplant.
  * Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL), Marginal Zone B-Cell Lymphoma, Follicular Lymphoma, which have progressed within 12 months of achieving a partial or complete remission. Patients who had remissions lasting > 12 months, are eligible after at least two prior therapies. Patients with bulky disease should be considered for debulking chemotherapy before transplant. Patients with refractory disease are eligible, unless has bulky disease and an estimated tumor doubling time of less than one month.
  * Lymphoplasmacytic Lymphoma, Mantle-Cell Lymphoma, Prolymphocytic Leukemia are eligible after initial therapy if chemotherapy sensitive.

Patients must have undergone an autologous transplant ≤ 12 months prior to allogeneic transplantation or have received multi-agent or immunosuppressive chemotherapy within 3 months of the preparative regimen.

* Adequate performance status defined as a Karnofsky score ≥ 70%
* Adequate organ function within 14 days (30 days for cardiac and pulmonary) of enrollment defined as:

  * Renal: creatinine < 2.0 mg/dL, for patient with a creatinine > 1.2 mg/dL or a history of renal dysfunction an estimated glomerular filtration rate > 40 mL/min/1.73 m2 is required
  * Hepatic: bilirubin, AST, ALT, alkaline phosphatase < 5 x upper limit of normal,
  * Pulmonary function: DLCOcorr > 40% normal,
  * Cardiac: left ventricular ejection fraction > 35%
* Voluntary written consent signed before performance of any study-related procedure not part of normal medical care

Exclusion Criteria:

* Untreated active infection at time of transplantation
* History of HIV infection
* Pregnant or breast feeding. The agents used in this study may be teratogenic to a fetus and there is no information on the excretion of agents into breast milk. Females of childbearing potential must have a blood test or urine study within 14 days prior to registration to rule out pregnancy
* Prior allogeneic transplantation
* Less than 3 months from myeloablative conditioning for autologous transplantation

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade II-IV acute graft-versus-host disease | Day +100
  Determine if 3:1 ratio of Treg:CD3+ cells reduces the risk grade II-IV acute graft versus host disease of 20% by day 100 as compared to patients with hematological malignancy receiving same conditioning regimen and immunosuppression but no Tregs.

SECONDARY OUTCOMES:
Incidence of double and single unit chimerism | Day +100
  Compare the incidence of double and single unit chimerism at day +100 between Treg and controls
Incidence of grade III-IV acute graft-versus-host disease | Day +100
  Compare the incidence of grade III-IV aGVHD between Treg and controls
Incidence of viral and fungal infections | 1 year
  Compare the incidence of viral and fungal infections at 1 year between Treg and controls
Survival | 1 year
  Compare the probability of survival at 1 year between Treg and controls
Incidence of neutrophil recovery | Day 42
  Compare the incidence of neutrophil recovery at day 42 between Treg and controls
Incidence of treatment related mortality | 6 months
  Determine the incidence of treatment related mortality (TRM) at 6 months between Treg and controls
Incidence of platelet recovery | 1 year
  Compare the incidence of platelet recovery at 1 year between Treg and controls
Incidence of chronic GVHD | 1 year
  Compare the incidence of chronic GVHD at 1 year between Treg and controls
Incidence of relapse | 1 year
  Compare the incidence of relapse at 1 year between Treg and controls

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Brunstein, MD, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota, United States